CLINICAL TRIAL: NCT04848116
Title: Neoadjuvant Targeting of Myeloid Cell Populations in Combination With Nivolumab in Head & Neck Cancer Patients Undergoing Surgery
Brief Title: Neoadjuvant Targeting of Myeloid Cell Populations in Combination With Nivolumab in Head & Neck Ca
Acronym: Spark2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J2085; IRB00254591 (Other: JHM IRB)
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; HuMax-IL8

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Nivolumab (240 mg) + HuMax/BMS-986253 (2400 mg) will be administered as an IV infusion.
  Interventions: Drug: Nivolumab; Drug: HuMax-IL8
- Cohort 2 (Experimental): Nivolumab (240 mg) + HuMax/BMS-986253 (3600 mg) will be administered as an IV infusion.
  Interventions: Drug: Nivolumab; Drug: HuMax-IL8

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is an investigational drug in this study.
  Other Names: BMS-936558
Drug: HuMax-IL8 — HuMax-IL8 is an investigational drug in this study.
  Other Names: BMS-986253

SUMMARY:
The primary objective of this study is to assess safety and feasibility of pre-operative nivolumab in combination with BMS-986253 (anti-interleukin-8) in patients with squamous cell carcinoma of head and neck (SCCHN) who will undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* The primary site should be a head and neck squamous cell carcinoma (including, but not limited to oral cavity, oropharynx, hypopharynx, or larynx, paranasal sinuses, nasal cavity). Squamous cell carcinoma of unknown primary, diagnosed in lymph nodes in neck, can be included but should be tested for p16 and confirmed with an HPV specific assay (testing NOT required for enrollment; can be done at an interval).
* Subjects must be human papillomavirus (HPV) negative (confirmed testing for oropharyngeal primary tumors - if otherwise suspected HPV positivity e.g. some oral cavity or sinonasal tumors if e.g. absence of smoking) OR (if HPV+) be high risk based on a ≥20 pack year smoking history.
* HPV testing is required per clinical standards
* Subjects must have been determined to be candidates for surgical resection by a multidisciplinary team including a surgeon, a medical oncologist and a radiation oncologist. Resection should typically be definitive but may also be done for symptomatic control e.g. in the setting of (suspected) metastatic disease with dominant local symptoms.
* Subjects must have at least one lesion that can be (or has been) biopsied at baseline.
* Patients with metastatic disease (both HPV(-) and high-risk HPV(+) (i.e. ≥20 pack years of smoking) are allowed, as long as patients have an indication for surgery for locoregional disease, and a life expectancy of ≥6 months. Metastatic disease can be addressed with additional treatments after trial treatment, e.g. focal radiation, or additional systemic therapy (e.g. chemotherapy or as indicated a targeted therapy or standard of care immunotherapy).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Age greater than or equal to 18 years
* Life expectancy of greater than 6 months
* Patients must have normal organ and marrow function
* The effects of nivolumab, as well as the other agents in this study on the developing human fetus are unknown.

  * Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
  * Women must not be breastfeeding
  * Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception as outlined in protocol
  * Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception as outlined in protocol
* Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated Institutional Review Board (IRB) approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report AEs, understand the drug dosing schedule and use of medications to control AEs
* Measurable disease - either radiologically (per RECIST) or clinically measurable on exam in order to assess treatment response.

Exclusion Criteria:

* Any active history of a known autoimmune disease. Subjects with vitiligo, type 1 diabetes mellitus, residual hypothyroidism requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Patients who received prior therapy with anti programmed death-1 (PD-1), anti-PD-L1, anti-PD-L2, anti CD137, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), anti-CSF1R, anti-interleukin-8 (IL8) therapies, any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Any live / attenuated vaccine (e.g. varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella (MMR) etc.) within 30 days of first dose of study treatment.
* Patients with uncontrolled brain metastases

Patients with brain metastases must have stable neurologic status following local therapy (surgery and/or radiation) for at least 2 weeks without the use of steroids or on stable or decreasing dose of ≤ 10mg daily prednisone (or equivalent), and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of carcinomatous meningitis are not eligible.

However, patients with metastatic disease (both HPV(-) and high-risk HPV(+) (i.e. ≥20 pack years of smoking) are allowed, as long as patients have an indication for surgery for locoregional disease, and a life expectancy for ≥6 months. Metastatic disease can be addressed with additional treatments after trial treatment, e.g. focal radiation, or additional systemic therapy (e.g. chemotherapy or as indicated a targeted therapy or standard of care immunotherapy).

* Patients who have an active concurrent malignancy that is not controlled/cured and could impact life expectancy within the next 3 years. E.g. patients with localized cutaneous squamous cell carcinoma or basal cell carcinoma or treated prostate cancer with no evidence of disease progression may be allowed to enroll after review by the study team and principal investigator.
* Uncontrolled inter-current illness including, but not limited to, no clinically significant active infection requiring (antimicrobial) treatment in the last week, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, myocardial infarction or new onset angina within six months of enrollment, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or nursing
* Men with female partners who are not willing to use contraception (Contraception method defined in protocol)
* Active infection with hepatitis B or hepatitis C (active infection is defined by either a) abnormal liver function tests (=elevated aspartate aminotransferase/alanine aminotransferase) or b) ongoing use of an antiviral hepatitis treatment).

  * Patients with normal liver function tests (=normal aspartate aminotransferase/alanine aminotransferase) and no antiviral medication per definition do not have an active infection and are eligible to enroll without additional testing).
  * Patients with normal liver function test do NOT need additional Hepatitis (no need for Hepatitis serology and/or PCR)
* Patients with a condition requiring chronic systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study start. However, inhaled or topical steroids and adrenal replacement steroid doses < 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Also, a burst of steroids (≤10 days use, e.g. a contrast premedication, or a methylprednisolone dose pack or similar) are acceptable and not excluded.
* Epstein-Barr Virus (EBV) positive head and neck cancer (e.g. EBV(+) nasopharyngeal carcinoma)
* Patients with HIV are excluded given the unknown risk of interaction with HAART and the unknown benefit of immunotherapy in this population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety of neoadjuvant Nivolumab in combination with HuMax | Up to 100 days after the last dose of study drug
  Adverse events will be reviewed to determine the safety of the combination of investigational products in the neoadjuvant setting. AEs and other toxicities will be graded using NCI Common Terminology Criteria for Adverse Events 5.0 (CTCAE).
Feasibility of neoadjuvant Nivolumab in combination with HuMax | Up to 100 days after the last dose of study drug
  Adverse events will be reviewed to determine the feasibility of the combination of investigational products in the neoadjuvant setting. AEs and other toxicities will be graded using NCI Common Terminology Criteria for Adverse Events 5.0 (CTCAE).

SECONDARY OUTCOMES:
Immune Related Pathologic Response | From neoadjuvant therapy to surgical resection, approximately 4 weeks
  Will be used to assess resection specimen and examine tumor regression.
Pathologic Response | From neoadjuvant therapy to surgical resection, approximately 4 weeks
  Examines total viable cells remaining after neoadjuvant therapy.
Relapse Free Survival | Up to 5 years after surgery
  The time measured between surgery and the development of signs/symptoms of cancer, if applicable.
Overall Survival | Up to 5 years after surgery
  Longevity of life after neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Fakhry, M.D., Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No